CLINICAL TRIAL: NCT02182505
Title: A Randomized, Double-blind Study to Compare the Safety and Efficacy of Berodual® Inhaled Via the Respimat® Device in Two Dosages (50 µg Fenoterol Hydrobromide + 20 µg Ipratropium Bromide and 25 µg Fenoterol Hydrobromide + 10 µg Ipratropium Bromide, 1 Puff t.i.d.) With That of Berodual® Inhaled Via the MDI With Aerochamber® (50 µg Fenoterol Hydrobromide + 21 µg Ipratropium Bromide, 2 Puffs t.i.d.) in Pediatric Patients With Asthma Over a 4 Week Period
Brief Title: Safety and Efficacy of Berodual® Inhaled Via Respimat® Compared to MDI (Metered Dose Inhaler) in Pediatric Patients With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 215.1105
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (3):
- Berodual® Respimat®, low dose (Experimental)
  Interventions: Drug: Berodual® Respimat®, low dose
- Berodual® Respimat®, high dose (Experimental)
  Interventions: Drug: Berodual® Respimat®, high dose
- Berodual® MDI Aerochamber® (Active Comparator)
  Interventions: Drug: Berodual® MDI

INTERVENTIONS:
Drug: Berodual® Respimat®, low dose
  Arms: Berodual® Respimat®, low dose
Drug: Berodual® Respimat®, high dose
  Arms: Berodual® Respimat®, high dose
Drug: Berodual® MDI
  Arms: Berodual® MDI Aerochamber®

SUMMARY:
Study to demonstrate that at least one of the two doses of Berodual® (50 µg fenoterol hydrobromide + 20 µg ipratropium bromide and 25 µg fenoterol hydrobromide + 10 µg ipratropium bromide, 1 puff t.i.d.) administered via Respimat® device gives a bronchodilator response which is not inferior to that obtained from one dose of Berodual® (50 µg fenoterol hydrobromide + 21 µg ipratropium bromide, 2 puffs t.i.d.) administered via the MDI (chlorofluorocarbon-metered dose inhaler) with Aerochamber® and that the safety profile is at least as good when paediatric asthma patients are treated for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bronchial asthma according to the ATS (American Thoracic Society) criteria
* Male or female children between 6 and 15 years old
* Screening FEV1: 60-90 % of predicted normal. Predicted normal values will be based on the reference values by Cotes
* Airway obstruction reversibility: FEV1 should increase ≥ 12% over baseline 30 to 60 minutes after administration of 2 puffs from the Berodual® MDI used with the Aerochamber®
* Ability to be trained in proper use of MDI with Aerochamber® and Respimat®
* Ability to perform technically satisfactory pulmonary function tests
* No hospital admission for an exacerbation and stable dosage of all pulmonary medication in the last four weeks
* Parent(s)/legal guardian is able and willing to give written informed consent in accordance with Good Clinical Practice (GCP) and local legislation. The child is willing to give oral consent

Exclusion Criteria:

* Patients with significant disease other than asthma, e.g. history of clinically significant cardiovascular, renal, neurological, hepatic or endocrine dysfunction (e.g. hyperthyreosis). A clinically significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or which may influence the results of the study or the ability of the patient to participate in and complete the study
* Tuberculosis with indication for treatment
* History of cancer within the last five years
* Patients who have undergone thoracotomy
* Current psychiatric disorders
* History of life threatening pulmonary obstruction, active bronchiectasis, lung fibrosis, AIDS (acquired immunity deficiency syndrome) and cystic fibrosis
* Severe bronchial asthma with frequent nocturnal asthma attacks or acute exacerbations induced by recurrent bronchial infections several times per year
* An upper or lower respiratory tract infection in the four weeks prior to the screening visit (= Visit 1) or during the 2-week run-in period
* Patients with known narrow-angle glaucoma or raised intra-ocular pressure
* Patients with known intolerance or hypersensitivity to any of the trial medication including excipients
* Patients using oral corticosteroid medication within the last 4 weeks
* Patients using leukotriene receptor antagonists and 5-LO (lipoxygenase) inhibitors within the last 4 weeks
* Beta-blocker medication
* Patients who have taken an investigational drug one month or six half-lives (whichever is greater) prior to the screening visit
* Previous participation in the run-in phase of this study
* Presence of psycho-social factors in the patient and/or relatives which, at the discretion of the investigator, do not assure compliance with medication, procedures and/or protocol

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 535 (Actual)
Dates: Start 1998-09; Primary Completion 1999-07 (Actual)

PRIMARY OUTCOMES:
Change in average FEV1 AUC0-1 (FEV1( (Forced expiratory volume in one second) AUC0-1(Area under the curve between 0 and 1 hour )) | pre-dose and 5, 30, 60 minutes post-dose on day 29

SECONDARY OUTCOMES:
Average FEV1 between 0 and 1 hour (FEV1 AUC0-1) | pre-dose and 5, 30, 60 minutes post-dose on days 1 and 15
Total average FEV1 between 0 and 1 hour (FEV1 AUC0-1) | pre-dose and 5, 30, 60 minutes post-dose on day 29
FVC (Forced vital capacity) | pre-dose and 5, 30, 60 minutes post-dose on days 1, 15 and 29
FEV25-75% (mean forced expiratory flow during the middle half of the FVC | pre-dose and 5, 30, 60 minutes post-dose on days 1, 15 and 29
FEV1max | pre-dose and 5, 30, 60 minutes post-dose on days 1 and 29
Onset of therapeutic response | Days 1 and 29
Peak expiratory flow (PEF) | pre-dose until day 29
Extent of use of rescue bronchodilator medication | up to day 29
Overall incidence of adverse events | up to day 29
Occurrence of application induced bronchoconstriction | up to day 29
Number of patients with clinically significant changes in heart rate | pre-dose and 5, 30, 60 minutes post-dose on days 1, 15, 29
Number of patients with clinically significant changes in blood pressure | pre-dose and 5, 30, 60 minutes post-dose on days 1, 15, 29
Number of patients with abnormal findings in physical examination | Baseline, day 29